CLINICAL TRIAL: NCT03565042
Title: Mechanism of Action Study of Ustekinumab Treatment in Psoriatic Arthritis: Impact on Cellular and Molecular Pathways of Synovial Inflammation and Tissue Remodeling
Brief Title: Mechanism of Action of Ustekinumab in Psoriatic Arthritis
Acronym: MoA anti-p40
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: Academisch Medisch Centrum - Universiteit van Amsterdam (AMC-UvA) (Other)
Responsible Party: Principal Investigator, D.L.P. Baeten, Prof. Dr. D.L.P. Baeten, Academisch Medisch Centrum - Universiteit van Amsterdam (AMC-UvA)
Other Study IDs: AMC_50218_MoA anti-p40
Record Dates: First submitted 2016-03-01; First posted 2018-06-21 (Actual); Last update posted 2018-06-21 (Actual); Status verified 2018-06

CONDITIONS: Arthritis, Psoriatic
Keywords: Arthritis, Psoriatic; Mechanism of Action; Ustekinumab; anti-p40; anti-IL23/Il12 p40
MeSH Terms: conditions — Arthritis, Psoriatic | interventions — Arthroscopy

STUDY DESIGN:
Observational Model: Other | Time Perspective: Prospective
Biospecimen Retention: Samples With DNA — * synovial tissue
  * synovial tissue both obtained at timepoint 0 (before first ustekinumab injection) ,wk 12, and wk24 after starting treatment
  * peripheral blood obtained at wk 0, wk 4, 8, 12 and 24
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (1):
- MoA ustekinumab: Patients with a diagnosis of psoriatic arthritis according to the CASPAR criteria with at least one swollen knee or ankle joint who are planning to receive treatment with ustekinumab at the outpatient clinic. An arthroscopy will be done in the swollen knee/ankle at week 0, 12 and 24.
  Interventions: Procedure: Arthroscopy

INTERVENTIONS:
Procedure: Arthroscopy — Arthroscopy of swollen joint (ankle/knee)

SUMMARY:
The purpose of this study is to determine the mechanism of action on target tissue level of ustekinumab treatment in psoriatic arthritis patients.

Patients who are planning to start treatment with anti-p40 therapy (ustekinumab) will be included in the trial.

At week 0, 12 and 24 peripheral blood, synovial tissue and skin will be obtained and analysed with different techniques to assess the effect of the therapy on inflammatory pathways.

DETAILED DESCRIPTION:
Rationale:

The overall aim of the study is to determine which downstream cellular and molecular pathways involved in psoriatic arthritis (PsA) pathogenesis are modulated by Interleukine 23/Interleukine12 P40 subunit (IL23/12 P40) blockade. As we have ample evidence that relevant disease-specific pathways are found in the primary target tissues, in particular in synovial tissue obtained from peripheral joints, but not in peripheral blood, we will strongly focus on this compartment by obtaining paired biopsies before and after treatment.

Objectives:

The primary objective is to assess the effect of IL23/12 P40 blockade on cellular en molecular pathways involved in PsA disease in the synovium, in the synovial fluid and peripheral blood.

The secondary objective is to compare which cellular/molecular disease pathways are affected by IL23/12 P40 blockade and not by tumour necrosis factor (TNF) blockade and thereby identify molecular biomarkers which may help to determine which patients may benefit from this treatment in comparison with anti-TNF treatment.

Study design:

Single centre, 24-week open-label study in subjects with clinically active peripheral psoriatic arthritis receiving treatment with ustekinumab.

Synovial biopsies will be obtained from patients before and after 12 and 24 weeks of treatment with ustekinumab.

Study population:

Patients with a diagnosis of psoriatic arthritis according to the Classification Criteria for Psoriatic Arthritis (CASPAR) criteria with at least one swollen knee or ankle joint who are planning to receive treatment with ustekinumab at the outpatient clinic. In total 16 patients will be included.

Intervention: Blood withdrawal and mini-arthroscopies at different timepoints.

Main study parameters/endpoints:

Primary study parameters/outcome of the study:

• Changes in the synovial cellular infiltrate and molecular pathways influenced between baseline and week 12/ week24

Secondary study parameters/outcome of the study:

• Comparison of the synovial molecular changes induced by anti-p40 with the changes induced by anti-TNF (analysed in historical samples in a similar patient population and study setting)

ELIGIBILITY:
Inclusion Criteria:

* Male and female patients age > 18 years diagnosed with Psoriatic Arthritis according to the CASPAR criteria
* Patient for whom the treating physician has decided to prescribe in the usual manner: Ustekinumab (Stelara) (45mg/ injection, given on week 0, 4, and every 12 weeks thereafter)
* Active disease defined by ≥1 swollen and ≥ 1 tender joint, and at least 1 swollen knee or ankle joint at baseline

Exclusion Criteria:

* Contraindications for needle-arthroscopy such as joint replacement (in the affected knee or ankle joint).
* Use of any investigational drug and/or devices within 4 weeks of baseline, or a period of 5 half-lives of the investigational drug, whichever is longer.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients with a diagnosis of psoriatic arthritis according to the CASPAR criteria with at least one swollen knee or ankle joint who are planning to receive treatment with ustekinumab at the outpatient clinic. In total 16 patients will be included.
Sampling Method: Non-Probability Sample
Enrollment: 16 (Estimated)
Dates: Start 2015-12-08 (Actual); Primary Completion 2018-10 (Estimated); Study Completion 2018-11 (Estimated)

PRIMARY OUTCOMES:
Biological effect of treatment on synovium obtained via arthroscopy from a swollen knee or ankle. | Cellular and molecular changes of the synovium of samples obtained at week 0 compared with week 12 and week 24.
  Cellular and molecular changes of the synovium.

OTHER OUTCOMES:
biological effect of anti TNF v.s. anti IL23/IL12 p40 on synovium obtained from a swollen knee or ankle. | week 0 compared with week 12 and week 24
  molecular and cellular changes affected by anti IL23/IL12 p40 and not by anit TNF therapy.

CONTACTS AND LOCATIONS:
Overall Officials: Dominique LP Baeten, MD PhD Prof, Principal Investigator — Academisch Medisch Centrum - Universiteit van Amsterdam (AMC-UvA)
Locations (1):
- Academic Medical Center Amsterdam, Amsterdam, North Holland, Netherlands